CLINICAL TRIAL: NCT02086396
Title: Effect of Hypoenergetic Diet Combined With Pumpkin Seed Flour Consumption on Obese Women
Brief Title: Effect of Weight Loss Diet and Pumpkin Seed Flour Consumption on Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Anna Paula Soares de Oliveira Carvalho, Masters in Cardiovascular Sciences, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACarvalho
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
Keywords: obesity; cardiovascular risk factors; pumpkin seed; diet quality
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pumpkin seed flour (Experimental): The pumpkin seed flour group received 20g/day of pumpkin seed flour during 12 weeks
  Interventions: Dietary Supplement: pumpkin seed flour
- Cassava flavored flour (Placebo Comparator): The placebo group (cassava flour flavored) received 20g/day of cassava flour flavored during 12 weeks.
  Interventions: Dietary Supplement: Placebo (cassava flavored flour)

INTERVENTIONS:
Dietary Supplement: pumpkin seed flour — The pumpkin seed flour group received 20g/day of pumpkin seed flour during 12 weeks
  Arms: pumpkin seed flour
Dietary Supplement: Placebo (cassava flavored flour) — The group placebo (cassava flour flavored) received 20g/day of cassava flour flavored during 12 weeks.
  Arms: Cassava flavored flour

SUMMARY:
This study aimed to evaluate the effect of weight loss diet combined with pumpkin seed flour consumption on diet improvement, weight loss, and glucose and cholesterol reduction in obese.

ELIGIBILITY:
Inclusion Criteria:

* age from 20 to 59 years old.
* body mass index above 30 kg/m2

Exclusion Criteria:

* diabetic
* loss weight before the research
* consumption of vitamins or dietary supplement.
* pregnancy

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Anthropometric measures | Change from Baseline at 12 weeks
  body weight (kg), body mass index (kg/m2), waist circumference (cm), neck circumference

SECONDARY OUTCOMES:
Blood lipids | Change from baseline at 12 weeks
  total Cholesterol (mg/dl), LDL-cholesterol (mg/dl), HDL-cholesterol (mg/dl) and triglycerides (mg/dl)
Blood glucose | Change from baseline at 12 weeks
  glucose (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Glorimar Rosa, Doctor, Study Director — Universidade Federal do Rio de Janeiro; Gláucia MM Oliveira, Doctor, Study Chair — Universidade Federal do Rio de Janeiro; Anna SO Carvalho, Master, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil